CLINICAL TRIAL: NCT01811472
Title: A Randomized, Multicenter, Double-blind, Placebo-controlled, Parallel-group, 24-week Pilot Study to Assess the Efficacy, Safety and Tolerability of LCQ908 in Patients With Non-alcoholic Fatty Liver Disease
Brief Title: Study to Assess the Efficacy, Safety and Tolerability of LCQ908 in NAFLD Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLCQ908A2216; 2013-000049-38 (EudraCT Number)
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD)
Keywords: Multi-center,; randomized,; double-blind,; NAFLD,; elevated triglycerides
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Hypertriglyceridemia | interventions — pradigastat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Patients randomized to Placebo arm, received matching placebo to 5 mg, 10 mg and 20 mg pradigstat (LCQ908) once daily for 24 weeks. Each patient was to receive 3 tablets a day. All patients were required to remain on their American Heart Association (AHA) diet for the entire duration of the study.
  Interventions: Drug: placebo
- pradigastat (LCQ908) 5mg/10mg (Experimental): Patients, randomized to pradigastat 5/10 mg, initially began with pradigastat (LCQ908) 5 mg once daily and then were up-titrated, if pradigastat (LCQ908) 5 mg once daily was tolerated, to pradigastat 10 mg once daily at Week 2. Total treatment duration was 24 weeks. Each patient was to receive 3 tablets a day. All patients were required to remain on their American Heart Association (AHA) diet for the entire duration of the study.
  Interventions: Drug: LCQ908
- pradigastat (LCQ908) 10mg/20mg (Experimental): Patients, randomized to pradigastat 10/20 mg, initially began with pradigastat (LCQ908) 10 mg once daily and then were up-titrated, if pradigastat (LCQ908) 10 mg once daily was tolerated, to pradigastat 20 mg once daily at Week 2. Total treatment duration was 24 weeks. Each patient was to receive 3 tablets a day. All patients were required to remain on their American Heart Association (AHA) diet for the entire duration of the study.
  Interventions: Drug: LCQ908

INTERVENTIONS:
Drug: LCQ908 — LCQ908 5 mg, 10 mg, 20 mg tablets
  Other Names: pradigastat
  Arms: pradigastat (LCQ908) 10mg/20mg; pradigastat (LCQ908) 5mg/10mg
Drug: placebo — Matching placebo of LCQ908 5 mg, 10 mg, 20 mg tablets.
  Arms: Placebo

SUMMARY:
The purpose of this study was to determine whether LCQ908 effectively lowers liver fat, as assessed by MRI and to assess its safety and tolerability profile in subjects with non-alcoholic fatty liver disease (NAFLD).

ELIGIBILITY:
Inclusion Criteria:

* History of liver steatosis during the preceding 24 months
* History of fasting TGs > 200 mg/dL (confirmed at screening).
* Liver fat ≥ 10% as determined by the central MRI laboratory.
* Subjects on the following medications can be included if these medications are medically necessary, cannot be stopped and the investigator feels their dose will remain stable for the duration of the double-blind treatment period:

  1. Stable dose of anti-diabetic medications (metformin and/or sulfonylureas) for at least 8 weeks prior to screening.
  2. Stable doses of beta-blockers and thiazide diuretics for at least 8 weeks prior to screening.
  3. Stable doses of fibrates, statins, niacin, ezetimibe for at least 8 weeks prior to screening.
  4. Stable dose of vitamin E in patients taking >200 IU/day for at least 6 months prior to screening.

Exclusion Criteria:

* Treatment with omega-3-acid ethyl esters or omega-3-polyunsaturated fatty acid (PUFA)-containing supplements > 200 mg per day within 8 weeks of screening.
* Treatment with antiretrovirals, tamoxifen, methotrexate, cyclophosphamide, isotretinoin, bile acid binding resins or pharmacologic doses of oral glucocorticoids (≥10 mg of prednisone per day or equivalent) within 8 weeks of screening.
* ALT or AST > 250 IU/L at the time of screening.
* History/current evidence of heavy alcohol use or alcoholism (> 21 drinks per week in men and > 14 drinks per week in women) over a 2-year period prior to screening.
* Presence of chronic liver disease, such as chronic hepatitis B and/or C, alcoholic liver disease, hemochromatosis, Wilson's disease, known cirrhosis.
* Platelet count <150,000 at screening.
* BMI >45 Kg/m2.

Other protocol defined inclusion/exclusion criteria may apply

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United States (11):
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Tamarac, Florida
  - Novartis Investigative Site, Honolulu, Hawaii
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Tupelo, Mississippi
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Plano, Texas
  - Novartis Investigative Site, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Pradigastat (LCQ908) 5mg/10mg | Pradigastat (LCQ908) 10mg/20mg
Started | 20 | 11 | 21
Completed | 18 | 11 | 16
Not Completed | 2 | 0 | 5
Not completed — Adverse Event | 1 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Subject/guardian decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included patients to whom study treatment was assigned excluding patients who were miss-randomized and did not take investigational drug. Mis-randomized patients were those who were not qualified for randomization, but were inadvertently randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pradigastat (LCQ908) 5mg/10mg | Pradigastat (LCQ908) 10mg/20mg | Total
Number analyzed (Participants) | 20 | 11 | 21 | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.9 (7.69) | 58.7 (6.56) | 47.7 (11.76) | 53.2 (10.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 10 | 26
  Male | 10 | 5 | 11 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Percentage of Fat in the Liver as Assessed Using MRI at Week 24
Description: Patients were to undergo MRI three times during the course of the study to assess liver fat. Baseline is defined as the value collected at Week -2 MRI assessment (approximately between Day -7 to -14).
Time Frame: From baseline to week 24
Population: Full analysis set included all patients to whom study treatment was assigned excluding patients who were miss-randomized and did not take investigational drug. Patients with baseline and post-baseline value at week 24 are included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of liver fat
Arm/Group | Placebo | Pradigastat (LCQ908) 5mg/10mg | Pradigastat (LCQ908) 10mg/20mg
Number analyzed (Participants) | 19 | 10 | 17
Percentage of liver fat | 0.00 [-1.63 to 1.63] | -1.68 [-3.93 to 0.56] | -2.89 [-4.59 to -1.18]
Statistical Analysis 1: Comparison: Placebo vs Pradigastat (LCQ908) 5mg/10mg; Hypothesis was tested at the 1-sided 5% significance level to assess if LCQ908 5mg/10mg was different from placebo; Test type: Non-Inferiority or Equivalence — The power calculation was largely driven by the maximum true response assumed in the candidate response shapes, which is a difference of -5.2% for pradigastat vs placebo for the primary endpoint; p = 0.3128, Mixed Model of Repeated Measurements; Degrees of freedom are adjusted using the Kenward-Roger method; Mean Difference (Net) = -1.69, 90% CI 2-sided [-4.46 to 1.09]
Statistical Analysis 2: Comparison: Placebo vs Pradigastat (LCQ908) 10mg/20mg; Hypothesis was tested at the 1-sided 5% significance level to assess if LCQ908 10mg/20mg was different from placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0457, Mixed Model of Repeated Measurements; Degrees of freedom are adjusted using the Kenward-Roger method; Mean Difference (Net) = -2.89, 90% CI 2-sided [-5.25 to -0.53]

2. Secondary Outcome: Change From Baseline in Percentage of Fat in the Liver as Assessed Using MRI at Week 12
Description: as for outcome 1
Time Frame: From baseline to week 12
Population: Full analysis set included all patients to whom study treatment was assigned excluding patients who were miss-randomized and did not take investigational drug. Patients with baseline and post-baseline value at week 12 are included in this analysis.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage of liver fat
Arm/Group | Placebo | Pradigastat (LCQ908) 5mg/10mg | Pradigastat (LCQ908) 10mg/20mg
Number analyzed (Participants) | 20 | 11 | 19
Percentage of liver fat | -0.80 [-2.31 to 0.72] | -1.71 [-3.79 to 0.37] | -2.98 [-4.55 to -1.42]

3. Secondary Outcome: Percentage of Responders at Week 12
Description: The response criteria are defined as:
  a. A reduction of ≥ 30% from baseline in liver fat b. A reduction of ≥ 50% from baseline in liver fat c. Liver fat content < 10% d. Liver fat content < 5.6%. Percentage is calculated as (m/n)*100 where m: number of patients who are responders. n: number of patients with non-missing percent liver fat at that visit.
Time Frame: At week 12
Population: Full analysis set included all patients to whom study treatment was assigned excluding patients who were miss-randomized and did not take investigational drug. Patients with non-missing percent liver fat at week 12 were included in this endpoint analysis.
Measure: Number; unit: Percentage of responders
Arm/Group | Placebo | Pradigastat (LCQ908) 5mg/10mg | Pradigastat (LCQ908) 10mg/20mg
Number analyzed (Participants) | 20 | 11 | 19
Percentage of responders
  At least 30% reduction in percent liver fat | 10.00 | 18.18 | 31.58
  At least 50% reduction in percent liver fat | 5.00 | 0.00 | 21.05
  Liver fat content < 10% | 5.00 | 18.18 | 36.84
  Liver fat content <5.6% | 0.00 | 0.00 | 21.05

4. Secondary Outcome: Percentage of Responders at Week 24
Description: as for outcome 3
Time Frame: From baseline to week 24
Population: Full analysis set included all patients to whom study treatment was assigned excluding patients who were miss-randomized and did not take investigational drug. Patients with non-missing percent liver fat at week 24 were included in this endpoint analysis.
Measure: Number; unit: Percentage of responders
Arm/Group | Placebo | Pradigastat (LCQ908) 5mg/10mg | Pradigastat (LCQ908) 10mg/20mg
Number analyzed (Participants) | 19 | 10 | 17
Percentage of responders
  At least 30% reduction in percent liver fat | 10.53 | 30.00 | 35.29
  At least 50% reduction in percent liver fat | 0.00 | 0.00 | 17.65
  Liver fat content < 10% | 5.26 | 20.00 | 52.94
  Liver fat content <5.6% | 0.00 | 0.00 | 17.65

5. Secondary Outcome: Change From Baseline Values for Alanine Aminotransferase (ALT) , Aspartate Aminotransferase (AST) and Gamma-glutamyl Transpeptidase (GGT) to Week 6
Description: Change from baseline ALT, AST and GGT values collected post-dose was analyzed using Mixed Model of Repeated Measurements (MMRM). Baseline is defined as the value collected at Week 0 (randomization).
  Treatment group and visit were fitted as factors and baseline was fitted as a continuous covariate.
Time Frame: From Baseline to week 6
Population: Full analysis set included all patients to whom study treatment was assigned excluding patients who were miss-randomized and did not take investigational drug. Patients with non-missing liver enzyme values at different timepoint were included in this endpoint analysis.
Measure: Least Squares Mean (90% Confidence Interval); unit: U/L
Arm/Group | Placebo | Pradigastat (LCQ908) 5mg/10mg | Pradigastat (LCQ908) 10mg/20mg
Number analyzed (Participants) | 20 | 11 | 20
U/L
  Liver enzyme: Alanine aminotransferase (ALT) | -2.6 [-10.6 to 5.3] | 1.4 [-9.2 to 12.1] | -9.1 [-17.0 to -1.1]
  Liver enzyme: Aspartate aminotransferase (AST) | 2.9 [-2.1 to 7.9] | 4.7 [-2.0 to 11.5] | -2.5 [-7.5 to 2.5]
  Liver enzyme: Gamma glutamyl transferase (GGT) | -13.9 [-22.1 to -5.7] | -7.0 [-18.1 to 4.0] | -0.9 [-9.1 to 7.3]

6. Secondary Outcome: Change From Baseline Values for Alanine Aminotransferase (ALT) , Aspartate Aminotransferase (AST) and Gamma-glutamyl Transpeptidase (GGT) to Week 12
Description: as for outcome 5
Time Frame: From Baseline to week 12
Population: Full analysis set included all patients to whom study treatment was assigned excluding patients who were miss-randomized and did not take investigational drug. Patients with non-missing liver enzyme values at week 12 were included in this endpoint analysis.
Measure: Least Squares Mean (90% Confidence Interval); unit: U/L
Arm/Group | Placebo | Pradigastat (LCQ908) 5mg/10mg | Pradigastat (LCQ908) 10mg/20mg
Number analyzed (Participants) | 20 | 11 | 20
U/L
  Liver enzyme: Alanine aminotransferase (ALT) | -0.6 [-10.3 to 9.1] | 2.9 [-10.2 to 16.0] | -3.7 [-13.8 to 6.4]
  Liver enzyme: Aspartate aminotransferase (AST) | 5.7 [-0.9 to 12.3] | 8.9 [0.0 to 17.7] | -0.1 [-7.1 to 6.9]
  Liver enzyme: Gamma glutamyl transferase (GGT) | -0.4 [-21.5 to 20.8] | -6.0 [-34.4 to 22.5] | 12.0 [-10.4 to 34.5]

7. Secondary Outcome: Change From Baseline Values for Alanine Aminotransferase (ALT) , Aspartate Aminotransferase (AST) and Gamma-glutamyl Transpeptidase (GGT) to Week 24
Description: as for outcome 5
Time Frame: From Baseline to week 24
Population: Full analysis set included all patients to whom study treatment was assigned excluding patients who were miss-randomized and did not take investigational drug. Patients with non-missing liver enzyme values at week 24 were included in this endpoint analysis.
Measure: Least Squares Mean (90% Confidence Interval); unit: U/L
Arm/Group | Placebo | Pradigastat (LCQ908) 5mg/10mg | Pradigastat (LCQ908) 10mg/20mg
Number analyzed (Participants) | 20 | 11 | 20
U/L
  Liver enzyme: Alanine aminotransferase (ALT) | -5.3 [-12.4 to 1.8] | -1.0 [-10.4 to 8.3] | -10.0 [-17.5 to -2.5]
  Liver enzyme: Aspartate aminotransferase (AST) | -1.8 [-7.9 to 4.3] | 2.5 [-5.4 to 10.4] | -3.2 [-9.6 to 3.3]
  Liver enzyme: Gamma glutamyl transferase (GGT) | -11.6 [-22.2 to -1.0] | -8.3 [-22.3 to 5.7] | 0.1 [-11.1 to 11.3]

8. Secondary Outcome: Percentage of Patients With Normalized Liver Enzymes
Description: Normalized liver enzymes defined as alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 40 U/L. Normal/High categories at baseline are defined by criteria of normal. Better is defined as high' at baseline and 'normal' post-dose; Same is defined as 'normal' at baseline and 'normal' post-dose or 'high' at baseline and 'high' post-dose; Worse is defined as 'normal' at baseline and 'high' post-dose.
Time Frame: Baseline, week 6, week 12 and week 24
Population: Full analysis set included all patients to whom study treatment was assigned excluding patients who were miss-randomized and did not take investigational drug. Patients with non-missing liver enzyme values at different timepoints were included in this endpoint analysis.
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | Pradigastat (LCQ908) 5mg/10mg | Pradigastat (LCQ908) 10mg/20mg
Number analyzed (Participants) | 20 | 11 | 20
Percentage of patients
  Better, week 6 | 10.0 | 0.0 | 10.0
  Same, week 6 | 85.0 | 90.9 | 85.0
  Worse, week 6 | 5.0 | 9.1 | 5.0
  Better, week 12 | 5.0 | 9.1 | 17.6
  Same, week 12 | 90.0 | 72.7 | 64.7
  Worse, week 12 | 5.0 | 18.2 | 17.6
  Better, week 24 | 5.3 | 18.2 | 17.6
  Same, week 24 | 89.5 | 72.7 | 58.8
  Worse, week 24 | 5.3 | 9.1 | 23.5

9. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides
Description: Blood samples were collected for a fasting triglycerides (TG) after a 10-hour (overnight) fast.
  Adjusted geometric means which is reported are calculated by back-transforming the adjusted means from the model and expressing as a percentage change from baseline. Baseline is defined as the value collected at Week 0 (randomization).
Time Frame: Baseline, 6, 12 and 24 weeks
Population: Full analysis set included all patients to whom study treatment was assigned excluding patients who were miss-randomized and did not take investigational drug. Patients with non-missing values at different timepoints were included in this endpoint analysis
Measure: Geometric Mean (90% Confidence Interval); unit: percent change
Arm/Group | Placebo | Pradigastat (LCQ908) 5mg/10mg | Pradigastat (LCQ908) 10mg/20mg
Number analyzed (Participants) | 20 | 11 | 21
percent change
  Change From Baseline to week 6 (n= 20,11, 20) | -14.6 [-26.5 to -0.8] | -16.0 [-31.3 to 2.8] | 3.2 [-11.1 to 19.8]
  Change From Baseline to week 12 (n = 20,11,17) | -7.3 [-18.2 to 5.2] | -7.9 [-22.3 to 9.1] | -15.8 [-26.5 to -3.5]
  Change From Baseline to week 24 (n= 19,11,17) | 13.0 [-3.8 to 32.6] | -10.0 [-27.3 to 11.3] | -2.4 [-17.6 to 15.5]

10. Secondary Outcome: Post-prandial Peak Triglycerides Over 0 - 8 Hours
Description: Post-prandial peak triglycerides is reported as maximum triglyceride value over 0-8 hours.
  Adjusted geometric means which is reported are calculated by back-transforming the adjusted means from the model. Baseline is defined as the value collected at Week 0 (randomization).
Time Frame: Baseline, 6 and 24 weeks
Population: as for outcome 9
Measure: Geometric Mean (90% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | Pradigastat (LCQ908) 5mg/10mg | Pradigastat (LCQ908) 10mg/20mg
Number analyzed (Participants) | 20 | 11 | 21
mg/dL
  Baseline (n= 20, 11, 21) | 394.0 [364.8 to 425.5] | 370.2 [333.8 to 410.6] | 375.9 [348.8 to 405.1]
  Week 6 (n = 20,11,20) | 336.0 [296.8 to 380.4] | 309.7 [262.1 to 366.0] | 374.1 [330.7 to 423.3]
  Week 24 (n= 20, 11, 15) | 401.5 [346.6 to 465.0] | 305.7 [205.9 to 372.5] | 351.8 [299.0 to 378.9]

11. Secondary Outcome: Change From Baseline in Body Weight
Time Frame: Baseline, 12 and 24 weeks
Population: Full analysis set included all patients to whom study treatment was assigned excluding patients who were miss-randomized and did not take investigational drug. Patients with both baseline and post-baseline values at different timepoints were included in this endpoint analysis
Measure: Least Squares Mean (90% Confidence Interval); unit: kilogram (kg)
Arm/Group | Placebo | Pradigastat (LCQ908) 5mg/10mg | Pradigastat (LCQ908) 10mg/20mg
Number analyzed (Participants) | 20 | 11 | 21
kilogram (kg)
  Change from baseline to week 12 (n=20, 11, 17) | -1.3 [-2.0 to -0.5] | -2.2 [-3.2 to -1.2] | -2.4 [-3.2 to -1.6]
  Change from baseline to week 24 (n=18, 11, 17) | -1.1 [-2.5 to 0.4] | -2.8 [-4.7 to -1.0] | -2.5 [-4.0 to -1.1]

12. Secondary Outcome: Change From Baseline in Waist Circumference
Time Frame: Baseline, 12 and 24 weeks
Population: as for outcome 11
Measure: Least Squares Mean (90% Confidence Interval); unit: centimeter (cm)
Arm/Group | Placebo | Pradigastat (LCQ908) 5mg/10mg | Pradigastat (LCQ908) 10mg/20mg
Number analyzed (Participants) | 20 | 11 | 21
centimeter (cm)
  Change from baseline to week 12 (n=20, 11, 17) | -0.4 [-2.3 to 1.6] | -3.7 [-6.4 to -1.0] | -4.2 [-6.3 to -2.1]
  Change from baseline to week 24 (n=19, 11, 17) | -1.7 [-3.9 to 0.6] | -3.7 [-6.7 to -0.6] | -4.2 [-6.6 to -1.9]

13. Secondary Outcome: Number of Patients With Adverse Events, Serious Adverse Events (SAEs) and Death as Assessment of Safety and Tolerability
Time Frame: 24 weeks
Population: Safety set (SAF) - All patients who received at least one dose of study drug and had at least 1 post-baseline safety assessment.
Measure: Number; unit: Patients
Arm/Group | Placebo | Pradigastat (LCQ908) 5mg/10mg | Pradigastat (LCQ908) 10mg/20mg
Number analyzed (Participants) | 20 | 11 | 21
Patients
  Patients with any adverse event | 14 | 9 | 20
  Patients with at least one SAE | 3 | 1 | 2
  Death | 0 | 0 | 0

ADVERSE EVENTS:
Description: Safety set (SAF) - All patients who received at least one dose of study drug and had at least 1 post-baseline safety assessment.
Groups:
- Pradigastat (LCQ908) 5mg /10 mg: Patients, randomized to pradigastat 5/10 mg, initially began with pradigastat (LCQ908) 5 mg once daily and then were up-titrated, if pradigastat (LCQ908) 5 mg once daily was tolerated, to pradigastat 10 mg once daily at Week 2. Total treatment duration was 24 weeks. Each patient was to receive 3 tablets a day. All patients were required to remain on their American Heart Association (AHA) diet for the entire duration of the study.
- Pradigastat (LCQ908) 10mg/20 mg: Patients, randomized to pradigastat 10/20 mg, initially began with pradigastat (LCQ908) 10 mg once daily and then were up-titrated, if pradigastat (LCQ908) 10 mg once daily was tolerated, to pradigastat 20 mg once daily at Week 2. Total treatment duration was 24 weeks. Each patient was to receive 3 tablets a day. All patients were required to remain on their American Heart Association (AHA) diet for the entire duration of the study.
- Pooled Pradigastat (LCQ908): This arm included all patients randomized to pradigastat (LCQ908) 5mg/10 mg and pradigastat (LCQ908)10mg/20 mg
Arm/Group | Placebo | Pradigastat (LCQ908) 5mg /10 mg | Pradigastat (LCQ908) 10mg/20 mg | Pooled Pradigastat (LCQ908)
Serious Adverse Events (participants affected / at risk) | 3/20 | 1/11 | 2/21 | 3/32
Other Adverse Events (participants affected / at risk) | 14/20 | 9/11 | 20/21 | 29/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=20) | Pradigastat (LCQ908) 5mg /10 mg (N=11) | Pradigastat (LCQ908) 10mg/20 mg (N=21) | Pooled Pradigastat (LCQ908) (N=32)
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 0 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
LUMBAR RADICULOPATHY (Nervous system disorders) | 1 | 0 | 0 | 0
SPINAL CLAUDICATION (Nervous system disorders) | 1 | 0 | 0 | 0
SYNCOPE (Nervous system disorders) | 0 | 0 | 1 | 1
DEPRESSION (Psychiatric disorders) | 0 | 0 | 1 | 1
PANIC ATTACK (Psychiatric disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=20) | Pradigastat (LCQ908) 5mg /10 mg (N=11) | Pradigastat (LCQ908) 10mg/20 mg (N=21) | Pooled Pradigastat (LCQ908) (N=32)
ANISOCYTOSIS (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
PALPITATIONS (Cardiac disorders) | 1 | 0 | 0 | 0
CONJUNCTIVITIS ALLERGIC (Eye disorders) | 1 | 0 | 0 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 | 0 | 0 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 3 | 2 | 3 | 5
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 | 1 | 10 | 11
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 1 | 2 | 3
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4 | 3 | 3 | 6
CONSTIPATION (Gastrointestinal disorders) | 4 | 0 | 3 | 3
DEFAECATION URGENCY (Gastrointestinal disorders) | 1 | 1 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 7 | 6 | 18 | 24
DYSPEPSIA (Gastrointestinal disorders) | 2 | 3 | 2 | 5
ERUCTATION (Gastrointestinal disorders) | 0 | 1 | 2 | 3
FAECES DISCOLOURED (Gastrointestinal disorders) | 0 | 1 | 0 | 1
FAECES HARD (Gastrointestinal disorders) | 2 | 1 | 0 | 1
FAECES SOFT (Gastrointestinal disorders) | 1 | 0 | 0 | 0
FLATULENCE (Gastrointestinal disorders) | 4 | 2 | 3 | 5
GASTROINTESTINAL MOTILITY DISORDER (Gastrointestinal disorders) | 3 | 1 | 0 | 1
GASTROINTESTINAL SOUNDS ABNORMAL (Gastrointestinal disorders) | 4 | 1 | 1 | 2
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 1 | 1 | 2
GINGIVAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 3 | 4 | 11 | 15
VOMITING (Gastrointestinal disorders) | 3 | 2 | 3 | 5
CHILLS (General disorders) | 0 | 0 | 2 | 2
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 0 | 0 | 0
BRONCHITIS (Infections and infestations) | 0 | 1 | 2 | 3
LYME DISEASE (Infections and infestations) | 0 | 1 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 4 | 2 | 0 | 2
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 | 1 | 0 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 1 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 2 | 0 | 2
URINARY TRACT INFECTION (Infections and infestations) | 0 | 2 | 0 | 2
CONTUSION (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
LACERATION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
STRESS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 0
RETICULOCYTE COUNT INCREASED (Investigations) | 0 | 1 | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 2
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 3
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 3
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
DIZZINESS (Nervous system disorders) | 2 | 1 | 1 | 2
HEADACHE (Nervous system disorders) | 1 | 4 | 1 | 5
HYPOAESTHESIA (Nervous system disorders) | 2 | 0 | 0 | 0
LUMBAR RADICULOPATHY (Nervous system disorders) | 0 | 1 | 0 | 1
MIGRAINE (Nervous system disorders) | 1 | 0 | 0 | 0
ANXIETY (Psychiatric disorders) | 1 | 0 | 2 | 2
INSOMNIA (Psychiatric disorders) | 0 | 0 | 2 | 2
HAEMATURIA (Renal and urinary disorders) | 0 | 1 | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1 | 0 | 1
URINE ODOUR ABNORMAL (Renal and urinary disorders) | 1 | 1 | 0 | 1
MENOPAUSAL SYMPTOMS (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 3
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.